CLINICAL TRIAL: NCT05150431
Title: Perioperative Pain-control With Parecoxib in Uniportal Video-assisted Thoracoscopic Surgery.
Brief Title: Optimized Acute Pain Control With Parecoxib in Uniportal Video-assisted Thoracoscopic Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202109025MINA
Record Dates: First submitted 2021-10-31; First posted 2021-12-09 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2021-10

CONDITIONS: Perioperative Care; Chronic Post-operative Pain
Keywords: Uniportal video-assisted thoracoscopy; enhanced recovery after surgery; parecoxib; chronic post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parecoxib (Experimental): Parecoxib 40mg will be administered to this group 15 minutes before the end of the surgery.
  Interventions: Drug: Parecoxib
- Placebo (Placebo Comparator): 2ml normal saline will be administered to this group 15 minutes before the end of the surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parecoxib — Parecoxib 40mg will be administered to the experimental group if the patient has no contraindication.
  Arms: Parecoxib
Drug: Placebo — This is normal saline 2ml, which is equal to the volume of parecoxib solution. Placebo will be injected to placebo group 15 minutes before the end of the surgery.
  Arms: Placebo

SUMMARY:
Chronic pain after thoracic surgery has been a bothering problem since the era of thoracotomy. The prevalence of chronic pain no matter in thoracotomy or video-assisted thoracoscopic surgery is about 30 to 47%. Better acute pain control after thoracic surgery has been assumed to be an effective way for prevention of chronic pain. Especially in this extreme minimal invasive surgery, uniportal video-assisted thoracic surgery, more optimized perioperative analgesics should be found out. In the guideline of "enhanced recovery after surgery", less opioid is suggested. Other than opioids, there are just few parental analgesics could be used, like acetaminophen or cyclooxygenase-2(COX-2) inhibitor. In our study, the investigators would like to build up a better analgesic strategy for uniportal video-assisted thoracoscopic surgery with less opioid and less side effects.

DETAILED DESCRIPTION:
Thoracic surgery has been progressed rapidly from traditional thoracotomy to triportal thoracoscopy, and even uniportal thoracoscopy within past decades. Perioperative pain control is always an important issue for postoperative recovery and prevention of chronic pain. The acute pain is most severe in the first 2 to 4 hours after the surgery until the chest tube removal. This painful sensation might postpone the ambulation time and restrain patient's respiratory depth or ability to cough. Although the surgical wound is getting smaller, the incidence of chronic pain is not declined as presumed. The incidence of chronic pain is highly related to acute pain control. In the guideline of enhanced recovery after lung surgery, multimodal analgesia is recommended. The combination of regional analgesia like thoracic epidural blockade (TEB) or paravertebral nerve blockade (PVB), and medications with different mechanism are beneficial for recovery. Intercostal nerve blockade is also studied and popular in recent years.

However, currently there is no optimal perioperative pain control suggestion for uniportal video-assisted thoracoscopic surgery (VATS). In uniportal VATS, the chest tube is the massive contribution for acute pain, and which is usually removed within postoperative 24 hours. In this study, the investigators would like to use the selective COX-2 inhibitor, parecoxib, combined with intra-operative intercostal nerve blockade for perioperative pain control. Parecoxib is relative long-acting than other currently using parental NSAID medication. The primary outcome is the morphine consumption in parecoxib and placebo groups. The secondary outcome is the numeric rating scale (NRS) during rest and cough, side effects, salvage medications, and chronic pain incidence in 3 months. The investigators hypothesized that parecoxib could effectively improve postoperative acute pain and reduce morphine consumption without serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled for uniportal video-assisted thoracoscopic surgery.
* The American Society of Anesthesiology (ASA) score is 1 or 2.

Exclusion Criteria:

* moderate to severe hepatic or renal insufficiency
* active peptic ulcer or gastrointestinal bleeding
* allergy to salicylates
* pregnancy or lactation period
* inflammatory bowel disease
* congestive heart failure
* accepted coronary artery bypass surgery
* ischemic heart disease
* peripheral vascular disease
* cerebrovascular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
post-operative 2-hour morphine consumption | 2 hours
  Patient-controlled analgesia will be provided to all the subjects in this study, immediately after the surgery. The investigators will record the total amounts of morphine consumption for each group.
post-operative 24-hour morphine consumption | 24 hours
  The investigators will record the given dosage of PCA in post-operative 24 hours.
post-operative 48-hour morphine consumption | 48 hours
  The investigators will record the given dosage of PCA in post-operative 48 hours.

SECONDARY OUTCOMES:
pain scale | 2 hours/24 hours/48 hours
  Resting and coughing numeric rating scale will be recorded for each group.
side effects caused by analgesics | 48 hours
  Dizziness, nausea, vomiting, voiding difficulty, respiratory depression will be recorded.
consumption of other analgesics, besides parecoxib and morphine | 24 hours/48 hours
  Additional salvage medication will be recorded and analyzed.
chronic pain prevalence | 3 to 6 months
  Telephone interview with a questionnaire will be used to follow the outcome of all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tzu Li, MD, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

REFERENCES:
- [Background] Mineo TC, Ambrogi V. A glance at the history of uniportal video-assisted thoracic surgery. J Vis Surg. 2017 Nov 7;3:157. doi: 10.21037/jovs.2017.10.11. eCollection 2017. PMID 29302433
- [Background] Gonzalez-Rivas D, Paradela M, Fernandez R, Delgado M, Fieira E, Mendez L, Velasco C, de la Torre M. Uniportal video-assisted thoracoscopic lobectomy: two years of experience. Ann Thorac Surg. 2013 Feb;95(2):426-32. doi: 10.1016/j.athoracsur.2012.10.070. Epub 2012 Dec 5. PMID 23219257
- [Background] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Background] Hazelrigg SR, Cetindag IB, Fullerton J. Acute and chronic pain syndromes after thoracic surgery. Surg Clin North Am. 2002 Aug;82(4):849-65. doi: 10.1016/s0039-6109(02)00031-2. PMID 12472133
- [Background] Tong Y, Wei P, Wang S, Sun Q, Cui Y, Ning N, Chen S, He X. Characteristics of Postoperative Pain After VATS and Pain-Related Factors: The Experience in National Cancer Center of China. J Pain Res. 2020 Jul 21;13:1861-1867. doi: 10.2147/JPR.S249134. eCollection 2020. PMID 32765060
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Turhan O, Sivrikoz N, Sungur Z, Duman S, Ozkan B, Senturk M. Thoracic Paravertebral Block Achieves Better Pain Control Than Erector Spinae Plane Block and Intercostal Nerve Block in Thoracoscopic Surgery: A Randomized Study. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):2920-2927. doi: 10.1053/j.jvca.2020.11.034. Epub 2020 Nov 20. PMID 33358107
- [Background] Maher DP, Wong W, White PF, McKenna R Jr, Rosner H, Shamloo B, Louy C, Wender R, Yumul R, Zhang V. Association of increased postoperative opioid administration with non-small-cell lung cancer recurrence: a retrospective analysis. Br J Anaesth. 2014 Jul;113 Suppl 1:i88-94. doi: 10.1093/bja/aeu192. Epub 2014 Jul 9. PMID 25009195
- [Background] Nussmeier NA, Whelton AA, Brown MT, Joshi GP, Langford RM, Singla NK, Boye ME, Verburg KM. Safety and efficacy of the cyclooxygenase-2 inhibitors parecoxib and valdecoxib after noncardiac surgery. Anesthesiology. 2006 Mar;104(3):518-26. doi: 10.1097/00000542-200603000-00020. PMID 16508400
- [Background] Shen H, Chen Y, Lu KZ, Chen J. Parecoxib for the prevention of shivering after general anesthesia. J Surg Res. 2015 Jul;197(1):139-44. doi: 10.1016/j.jss.2015.03.011. Epub 2015 Mar 28. PMID 25908099
- [Background] Huang JM, Lv ZT, Zhang B, Jiang WX, Nie MB. Intravenous parecoxib for early postoperative cognitive dysfunction in elderly patients: evidence from a meta-analysis. Expert Rev Clin Pharmacol. 2020 Apr;13(4):451-460. doi: 10.1080/17512433.2020.1732815. Epub 2020 Feb 28. PMID 32077347
- [Background] Bian YY, Wang LC, Qian WW, Lin J, Jin J, Peng HM, Weng XS. Role of Parecoxib Sodium in the Multimodal Analgesia after Total Knee Arthroplasty: A Randomized Double-blinded Controlled Trial. Orthop Surg. 2018 Nov;10(4):321-327. doi: 10.1111/os.12410. PMID 30485685